CLINICAL TRIAL: NCT01798706
Title: A Randomized, Double-blind, Placebo-controlled, 2-arm Parallel-group, Multicenter, 24 Week Study Assessing the Safety and Efficacy of Lixisenatide in Older Patients With Type 2 Diabetes Inadequately Controlled on Their Current Diabetes Treatment Regimen
Brief Title: Efficacy and Safety of Lixisenatide Versus Placebo on Top of Basal Insulin and/or Oral Antidiabetic Treatment in Older Type 2 Diabetic Patients
Acronym: GetGoal-O
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC12703; 2012-003292-19 (EudraCT Number); U1111-1132-9156 (Other: UTN)
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): Lixisenatide 10 mcg once daily (QD) for 2 weeks, then at a maintenance dose of 20 mcg QD up to Week 24. If the maintenance dose of 20 mcg was not tolerated, dose could be reduced to 10 mcg.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Antidiabetic background therapy
- Placebo (Placebo Comparator): Placebo (matched to lixisenatide) QD for 24 Weeks.
  Interventions: Drug: Placebo; Drug: Antidiabetic background therapy

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: Solution for injection in pre-filled pen administered 30 to 60 minutes before breakfast in the morning
  Route of administration: Subcutaneous injection
  Other Names: Lyxumia
  Arms: Lixisenatide
Drug: Placebo — Pharmaceutical form: Solution for injection in pre-filled pen administered 30 to 60 minutes before breakfast in the morning
  Route of administration: Subcutaneous injection
  Arms: Placebo
Drug: Antidiabetic background therapy — Participants received a stable regimen of anti-diabetic background therapy for at least 3 months prior to screening, during the placebo run-in period and the 24 week treatment period. Allowed background antidiabetic therapy included metformin, sulfonylurea (except glibenclamide >10 mg, gliclazide >160 mg), meglitinides (except repaglinide >6 mg), pioglitazone and basal insulin. Insulin glargine, neutral protamine hagedorn (NPH) insulin, detemir, lente and ultralente were considered as basal insulin.

SUMMARY:
Primary objective:

- To evaluate the effect of lixisenatide versus placebo over a period of 24 weeks on glycemic control, as evaluated by glycosylated hemoglobin (HbA1c) reduction, in older type 2 diabetes participants (T2DM) who are inadequately controlled with their current anti-diabetic treatment regimen.

Main secondary objective:

- To assess the safety and tolerability of lixisenatide compared to placebo in older T2DM participants (including occurrence of documented (Plasma Glucose PG < 60 mg/dL) symptomatic hypoglycemia and gastrointestinal side effects).

Other secondary objectives:

* To assess the effect of lixisenatide compared to placebo after 24-week treatment on:

  * Fasting plasma glucose (FPG);
  * During liquid standardized breakfast meal challenge test : 2 hour- Postprandial Plasma Glucose (PPG) and Plasma Glucose Excursion;
  * 7-point Self-monitored plasma glucose (SMPG) profile;
  * Body weight;
  * Change in total daily dose of basal insulin (if taken);
  * Percentage of participants requiring rescue therapy
  * Safety and tolerability;
* To assess lixisenatide pharmacokinetic profile;
* To assess anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
Approximately 31 weeks including 24 week treatment period.

ELIGIBILITY:
Inclusion criteria :

* Older participants, aged 70 years and above, with T2DM inadequately controlled on their current anti-diabetic pharmaceutical treatment regimen.
* Signed written informed consent.

Exclusion criteria:

* At screening HbA1c ≤7.0% or >10% (Acknowledging that the threshold of 7% may not be appropriate for all older participants and that this was the responsibility of the investigator to include the participant based on an individual evaluation of the expected benefits of better glycemic control versus risk of hypoglycemia).
* At screening participants on both basal insulin and sulfonylurea or basal insulin and meglitinides.
* At screening FPG >250 mg/dL (>13.9 mmol/L).
* Type 1 diabetes mellitus or history of ketoacidosis within one year prior to the screening visit.
* Type 2 diabetes mellitus diagnosed less than 1 year prior to screening.
* Anti-diabetic treatment not at a stable regimen or initiated within the last 3 months prior to screening.
* Treatment within the 3 months preceding the screening with other anti-diabetic agent than allowed background therapy. Allowed therapy includes metformin, sulfonylurea (except glibenclamide >10mg, gliclazide >160mg), meglitinides (except repaglinide >6mg), pioglitazone and basal insulin and should follow local product circulars and labeling restrictions for the study population.
* Participants who had been on an approved or an investigational Glucagon-like peptide 1 (GLP-1) medication (exenatide, liraglutide, lixisenatide or others).
* History of severe hypoglycemia associated with symptoms unawareness or results in unconsciousness/coma/seizure in the 6 months prior to screening.
* BMI <22 or >40 kg/m^2.
* Malnutrition assessed clinically by the investigator or any sub-investigator and by Mini-Nutritional Assessment-Short Form (MNA-SF) score <12 in countries (the judgment of the investigator prevails on questionnaires scores).
* Cognitive disorder and dementia assessed clinically by the investigator or any sub investigator and by Mini Mental State Examination (MMSE) score <24 (the judgment of the investigator prevails on questionnaires scores), or any neurologic disorder that affected the participant's ability to participate in the study.
* Participant who had a glomerular filtration rate (eGFR) (using the Modification of Diet in Renal Disease (MDRD) formula <30ml/min/1.73m^2).
* Participant with severe or uncontrolled disease, or any clinically significant abnormality identified on physical examination or investigational clinical procedure that, in the judgment of the investigator or any sub-investigator, would preclude safe completion of the study or constrains efficacy assessment.
* Laboratory findings at the time of screening:

  * Amylase and/or lipase: >3 times the upper limit of the normal (ULN) laboratory range
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times ULN
  * Calcitonin >20 pg/mL (5.9 pmol/L).
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (i.e. worsening) and not controlled (i.e. prolonged nausea and vomiting) gastroesophageal reflux disease within 6 months prior to screening.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease.
* Personal or immediate family history of medullary thyroid cancer or genetic conditions that predisposed to medullary thyroid cancer (e.g., multiple endocrine neoplasia syndromes).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 350 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (83):
- United States (14):
  - Investigational Site Number 840010, La Jolla, California
  - Investigational Site Number 840015, Norwalk, California
  - Investigational Site Number 840003, Miami, Florida
  - Investigational Site Number 840012, Miami, Florida
  - Investigational Site Number 840002, Des Moines, Iowa
  - Investigational Site Number 840008, Oxon Hill, Maryland
  - Investigational Site Number 840004, Rockville, Maryland
  - Investigational Site Number 840017, Biloxi, Mississippi
  - Investigational Site Number 840009, Omaha, Nebraska
  - Investigational Site Number 840016, Salisbury, North Carolina
  - Investigational Site Number 840006, Fargo, North Dakota
  - Investigational Site Number 840014, Canal Fulton, Ohio
  - Investigational Site Number 840011, St. George, Utah
  - Investigational Site Number 840007, Milwaukee, Wisconsin
- Australia (6):
  - Investigational Site Number 036002, Box Hill
  - Investigational Site Number 036006, Brookvale
  - Investigational Site Number 036004, Camperdown
  - Investigational Site Number 036005, Gosford
  - Investigational Site Number 036001, Heidelberg
  - Investigational Site Number 036003, Parkville
- Bulgaria (5):
  - Investigational Site Number 100002, Plovdiv
  - Investigational Site Number 100005, Plovdiv
  - Investigational Site Number 100003, Sofia
  - Investigational Site Number 100004, Stara Zagora
  - Investigational Site Number 100001, Varna
- Canada (8):
  - Investigational Site Number 124003, Hamilton
  - Investigational Site Number 124007, London
  - Investigational Site Number 124001, Saint Romuald
  - Investigational Site Number 124002, Sherbrooke
  - Investigational Site Number 124005, Vancouver
  - Investigational Site Number 124006, Vancouver
  - Investigational Site Number 124008, Westmount
  - Investigational Site Number 124004, Winnipeg
- Denmark (5):
  - Investigational Site Number 208005, Esbjerg
  - Investigational Site Number 208001, København NV
  - Investigational Site Number 208004, København S
  - Investigational Site Number 208002, Slagelse
  - Investigational Site Number 208003, Svendborg
- Germany (8):
  - Investigational Site Number 276005, Dresden
  - Investigational Site Number 276004, Essen
  - Investigational Site Number 276002, München
  - Investigational Site Number 276001, Münster
  - Investigational Site Number 276006, Pirna
  - Investigational Site Number 276007, Pohlheim
  - Investigational Site Number 276008, Potsdam
  - Investigational Site Number 276003, Saarlouis
- Norway (5):
  - Investigational Site Number 578001, Hønefoss
  - Investigational Site Number 578005, Kongsvinger
  - Investigational Site Number 578003, Oslo
  - Investigational Site Number 578006, Stavanger
  - Investigational Site Number 578004, Trondheim
- Peru (8):
  - Investigational Site Number 604001, Arequipa
  - Investigational Site Number 604011, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604003, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604002, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604008, Piura
- Poland (5):
  - Investigational Site Number 616004, Gdansk
  - Investigational Site Number 616003, Krakow
  - Investigational Site Number 616001, Poznan
  - Investigational Site Number 616002, Ruda Śląska
  - Investigational Site Number 616006, Szczecin
- South Africa (3):
  - Investigational Site Number 710003, Cape Town
  - Investigational Site Number 710002, Cape Town
  - Investigational Site Number 710004, Somerset West
- Spain (6):
  - Investigational Site Number 724001, Alzira
  - Investigational Site Number 724005, Barcelona
  - Investigational Site Number 724006, Hostalets de Balenyà
  - Investigational Site Number 724003, Madrid
  - Investigational Site Number 724002, Sanlúcar de Barrameda
  - Investigational Site Number 724004, Santiago de Compostela
- Sweden (6):
  - Investigational Site Number 752006, Gothenburg
  - Investigational Site Number 752007, Härnösand
  - Investigational Site Number 752002, Lund
  - Investigational Site Number 752004, Malmo
  - Investigational Site Number 752003, Stockholm
  - Investigational Site Number 752001, Stockholm
- United Kingdom (4):
  - Investigational Site Number 826003, Bexhill-on-Sea
  - Investigational Site Number 826001, Glasgow
  - Investigational Site Number 826002, Irvine
  - Investigational Site Number 826004, Trowbridge

REFERENCES:
- [Result] Meneilly GS, Roy-Duval C, Alawi H, Dailey G, Bellido D, Trescoli C, Manrique Hurtado H, Guo H, Pilorget V, Perfetti R, Simpson H; GetGoal-O Trial Investigators. Lixisenatide Therapy in Older Patients With Type 2 Diabetes Inadequately Controlled on Their Current Antidiabetic Treatment: The GetGoal-O Randomized Trial. Diabetes Care. 2017 Apr;40(4):485-493. doi: 10.2337/dc16-2143. Epub 2017 Feb 10. PMID 28188240
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 83 centers in 13 countries. A total of 786 participants were screened between June 10, 2013 and July 09, 2014.
Pre-assignment Details: A total of 426 participants underwent 4 week placebo run-in period. 436 participants were screen failures and 76 were run-in failures; the most frequent reason for screen and run-in failure was glycosylated hemoglobin (HbA1c) criteria not met at end of the run-in phase. A total of 350 participants were randomized.
Groups:
- Lixisenatide: Lixisenatide 10 mcg subcutaneously once daily (QD) for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to Week 24. If the maintenance dose of 20 mcg was not tolerated, dose could be reduced to 10 mcg.
- Placebo: Placebo (matched to lixisenatide) subcutaneously QD for 24 Weeks.
Period: Overall Study
Arm/Group | Lixisenatide | Placebo
Started | 176 | 174
Completed | 155 | 153
Not Completed | 21 | 21
Not completed — Adverse Event | 15 | 10
Not completed — Lack of Efficacy | 0 | 2
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Other than specified above | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Lixisenatide: Lixisenatide 10 mcg subcutaneously QD for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to Week 24. If the maintenance dose of 20 mcg was not tolerated, dose could be reduced to 10 mcg.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide | Placebo | Total
Number analyzed (Participants) | 176 | 174 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (4) | 74.4 (3.8) | 74.2 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 84 | 168
  Male | 92 | 90 | 182
Race [Number; unit: participants]
  Caucasian/white | 128 | 122 | 250
  Black | 3 | 0 | 3
  Asian/Oriental | 5 | 11 | 16
  Other | 40 | 41 | 81
Ethnicity [Number; unit: participants]
  Hispanic | 51 | 48 | 99
  Not Hispanic | 125 | 126 | 251
Number of Participants with Categorical BMI [Number; unit: participants]
  <30 kg/m^2 | 102 | 96 | 198
  ≥30 kg/m^2 | 74 | 78 | 152
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.91 (3.7) | 30.09 (4.53) | 30.00 (4.13)
Body Weight [Mean (Standard Deviation); unit: kg] | 80.81 (14.54) | 80.08 (16.76) | 80.45 (15.66)
HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.04 (0.72) | 8.05 (0.69) | 8.04 (0.71)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.83 (2.38) | 8.89 (2.26) | 8.86 (2.32)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — 347 participants (174 in lixisenatide arm and 173 in placebo arm) were included for PPG analysis.
  mmol/L | 15.18 (3.78) | 14.87 (3.69) | 15.03 (3.74)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — 345 participants (173 in lixisenatide arm and 172 in placebo arm) were included for glucose excursion analysis.
  mmol/L | 6.51 (3.15) | 6.02 (3.17) | 6.26 (3.16)
7-Point Self-monitored Plasma Glucose (SMPG) [Mean (Standard Deviation); unit: mmol/L] — 333 participants (171 in lixisenatide arm and 162 in placebo arm) were included for 7 point SMPG analysis.
  mmol/L | 9.79 (2.02) | 9.97 (1.98) | 9.87 (2.00)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 13.63 (7.34) | 14.63 (7.87) | 14.13 (7.62)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in HbA1c From Baseline to Week 24
Description: Change in HbA1c was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using last on-treatment observation carried forward (LOCF). On-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. Here, number of participants analyzed=participants with baseline and at least one post-baseline HbA1c assessment during on-treatment period.
Time Frame: Baseline, Week 24
Population: Modified intent to treat (mITT) population: all randomized participants who received at least one dose of study drug; and had both baseline and at least one post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 172 | 172
percentage of hemoglobin | -0.57 (0.075) | 0.06 (0.072)
Statistical Analysis 1: Comparison: Lixisenatide vs Placebo; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of basal insulin use at screening, randomization strata of Week -1 glomerular filtration rate (eGFR) (≥30 to <60, ≥60 ml/min/1.73 m^2), and country as fixed effects and baseline HbA1c value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -0.64, 95% CI 2-sided [-0.81 to -0.464], Standard Error of Mean 0.088 — Lixisenatide vs Placebo

2. Secondary Outcome: Change in 2-Hour PPG From Baseline to Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a liquid standardized breakfast meal. Change in PPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed=participants with baseline and at least one post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 147 | 144
mmol/L | -5.12 (0.392) | -0.07 (0.393)
Statistical Analysis 1: Comparison: Lixisenatide vs Placebo; Analysis was performed using ANCOVA model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of basal insulin use at screening, randomization strata of Week -1 eGFR (≥30 to <60, ≥60 ml/min/1.73 m^2), and country as fixed effects and baseline 2-hour PPG value as a covariate. Hierarchical testing procedure was used to control type I error at 0.05. Testing was then performed sequentially in the order the endpoints were reported; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level. Testing sequence continued only when previous endpoint was statistically significant at 0.05; LS Mean Difference = -5.05, 95% CI 2-sided [-5.96 to -4.132], Standard Error of Mean 0.464 — Lixisenatide vs Placebo

3. Secondary Outcome: Change in Average 7-point SMPG Profiles From Baseline to Week 24
Description: Participants recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime three times in a week before baseline, before visit Week 12 and before visit week 26 and the average value across the profiles performed in the week a visit for the 7-time points was calculated. Change in average 7-point SMPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed=participants with baseline and at least one post-baseline 7-point SMPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 138 | 125
mmol/L | -1.15 (0.186) | -0.19 (0.189)
Statistical Analysis 1: Comparison: Lixisenatide vs Placebo; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of basal insulin use at screening, randomization strata of Week -1 eGFR (≥30 to <60, ≥60 ml/min/1.73 m^2), and country as fixed effects and baseline 7-point SMPG value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.96, 95% CI 2-sided [-1.39 to -0.527], Standard Error of Mean 0.219 — Lixisenatide vs Placebo

4. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug up to 3 days after the last dose of study drug.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed=participants with baseline and at least one post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 174 | 173
kg | -1.47 (0.241) | -0.16 (0.228)
Statistical Analysis 1: Comparison: Lixisenatide vs Placebo; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of basal insulin use at screening, randomization strata of Week -1 eGFR (≥30 to <60, ≥60 ml/min/1.73 m^2), and country as fixed effects and baseline body weight value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -1.32, 95% CI 2-sided [-1.862 to -0.769], Standard Error of Mean 0.278 — Lixisenatide vs Placebo

5. Secondary Outcome: Change in FPG From Baseline to Week 24
Description: Change in FPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to 1 day after the last dose of study drug.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed=participants with baseline and at least one post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 171 | 168
mmol/L | -0.3 (0.224) | 0.01 (0.218)
Statistical Analysis 1: Comparison: Lixisenatide vs Placebo; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of basal insulin use at screening, randomization strata of Week -1 eGFR (≥30 to <60, ≥60 ml/min/1.73 m^2), and country as fixed effects and baseline FPG value as a covariate; Test type: Superiority or Other; p = 0.2347, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.31, 95% CI 2-sided [-0.828 to 0.204], Standard Error of Mean 0.262 — Lixisenatide vs Placebo

6. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy During 24 Week Treatment Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after Week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after Week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 mg/dL (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >9%.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 175 | 173
percentage of participants | 2.9 | 10.4

7. Secondary Outcome: Change in Plasma Glucose Excursions From Baseline to Week 24
Description: Plasma glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the liquid standardized breakfast meal test, before study drug administration. Change in plasma glucose excursions were calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants=participants with baseline and at least one post-baseline plasma glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 145 | 143
mmol/L | -4.71 (0.331) | -0.25 (0.331)

8. Secondary Outcome: Change in Total Daily Basal Insulin Dose From Baseline to Week 24 (in Participants Who Took Basal Insulin as Background Therapy)
Description: Change in basal insulin dose was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. The on-treatment period for this efficacy variable was the time from the first dose of study drug up to the day of last dose of study drug.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed=participants with baseline and at least one post-baseline basal insulin dose assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: units
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 54 | 55
units | -2.97 (1.145) | -1.3 (1.076)

9. Secondary Outcome: Percentage of Participants With Symptomatic and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the participant required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration (maximum of 171 days)
Population: Analysis was performed on safety population defined as all randomized participants who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 176 | 174
percentage of participants
  Symptomatic hypoglycemia | 7.4 | 5.7
  Severe symptomatic hypoglycemia | 0.57 | 0

10. Secondary Outcome: Percentage of Participants With HbA1c Reduction >0.5% at Week 24 and Did Not Experienced Documented (Plasma Glucose <60 mg/dL) Symptomatic Hypoglycemia
Description: The on-treatment period for HbA1c assessment was defined as the time from the first dose of study drug up to 14 days after the last dose of study drug. The on-treatment period for symptomatic hypoglycemia assessment was defined as the time from the first dose of study drug up to 1 day after the last dose of study drug.
Time Frame: Week 24
Population: mITT population. Participants without any post-baseline on-treatment value for HbA1c were counted as non-responders if they experienced at least one symptomatic hypoglycemia. Otherwise, they were counted as missing.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 172 | 172
percentage of participants | 57.6 | 21.5

11. Secondary Outcome: Percentage of Participants With Gastrointestinal Disorders
Time Frame: Up to Day 171
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Lixisenatide | Placebo
Number analyzed (Participants) | 176 | 174
percentage of participants | 40.3 | 20.7

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from signature of the informed consent form up to the final visit (Day 171) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the first dose of study drug up to 3 days after the last dose of study drug).
Groups:
- Lixisenatide: Lixisenatide 10 mcg subcutaneously QD for 2 weeks post-randomization, then at a maintenance dose of 20 mcg QD up to Week 24. If the maintenance dose of 20 mcg was not tolerated, dose could be reduced to 10 mcg.(Median exposure: 169 days)
- Placebo: Placebo (matched to lixisenatide) subcutaneously QD for 24 Weeks. (Median exposure: 169 days)
Arm/Group | Lixisenatide | Placebo
Serious Adverse Events (participants affected / at risk) | 8/176 | 10/174
Other Adverse Events (participants affected / at risk) | 89/176 | 58/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=176) | Placebo (N=174)
Bronchitis (Infections and infestations) | 0 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide (N=176) | Placebo (N=174)
Diarrhoea (Gastrointestinal disorders) | 19 | 13
Nausea (Gastrointestinal disorders) | 44 | 13
Vomiting (Gastrointestinal disorders) | 10 | 1
Nasopharyngitis (Infections and infestations) | 15 | 22
Hypoglycaemia (Metabolism and nutrition disorders) | 30 | 18
Headache (Nervous system disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.